CLINICAL TRIAL: NCT06453707
Title: Sample Type Validation: Finger Prick and Plasma vs Whole Blood in a Clinical Setting for the SpinChip High-sensitivity Cardiac Troponin I (SpinChip Hs-cTnI) Test
Brief Title: SpinChip Hs-cTnI Sample Type Validation
Acronym: HEAT-2
Status: Completed | Type: Observational
Sponsor: SpinChip Diagnostics ASA (Industry)
Collaborators: Aurevia (Industry); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Other Study IDs: Design Protocol-03645; CIV-NO-24-01-045754 (Other: EUDAMED)
Record Dates: First submitted 2024-05-29; First posted 2024-06-12 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; High-sensitive; Point of Care; Troponin I; Near-patient test; Heart attack
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Li-heparin plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SpinChip hs-cTnI — SpinChip Platform, consisting of the SpinChip hs-cTnI test (self-contained cartridge) and SpinChip Analyzer (instrument)

SUMMARY:
During a heart attack, the protein troponin I is released from the heart muscle into the bloodstream. Measurements of cardiac troponin in blood are used as an aid in the diagnosis of heart attack. The SpinChip hs-cTnI test is a new high-sensitive test for measuring the amount of cardiac troponin I in the bloodstream as an aid in the diagnosis of heart attack.

The purpose of this study is to demonstrate that different types of blood samples (finger prick, venous whole blood and plasma) return comparable results when analysed using the SpinChip hs-cTnI test. Blood samples from at least 150 patients will be analyzed and the testing will be carried out by healthcare personnel.

DETAILED DESCRIPTION:
Cardiac troponins are widely used as a biomarker to aid in the diagnosis of Acute myocardial infarction (AMI). These structural proteins are essential in regulating contraction in cardiac muscle cells, and they are sensitive and specific biochemical markers of myocardial damage.

During a heart attack, cardiac muscle cells are injured and release the cardiac marker troponin I (cTnI) into the bloodstream. High-sensitive troponin tests may detect the increase of cardiac troponin in blood within hours after the symptoms of a heart attack has started.

The SpinChip high-sensitivity cardiac troponin I (hs-cTnI) test is a new high-sensitive test for measuring troponin I in blood samples, and the analysis may be performed close to the patient (near-patient test). The results may be obtained within 10 minutes, compared to approximately 1 hour for normal laboratory analysis.

The SpinChip Platform consists of the SpinChip hs-cTnI test and the SpinChip Analyzer and may be used at the emergency department to evaluate patients presenting with symptoms of acute myocardial infarction (chest pain). The test can use blood from finger prick or venous blood samples, either as whole blood or separated into plasma.

The purpose of this study is to demonstrate that different sample types (finger prick, venous whole blood or plasma) give comparable results when analysed using the SpinChip hs-cTnI test when the testing is performed by healthcare professionals. Samples from minimum 150 patients with troponin levels covering the measuring range of the SpinChip hs-cTnI test will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed written informed consent
* Subjects >18 years old
* Clinical cardiac Troponin T concentration available

Exclusion Criteria:

* Cognitive impairment precluding informed consent
* Self-reported pregnancy
* General clinical condition which affects the patient in a major way and the patient is considered to be in an unstable clinical condition
* Previously included in the study with a sample within the measuring range of the SpinChip hs-cTnI test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minimum 150 hospitalized patients identified based on cardiac troponin levels obtained from clinical records at Akershus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Sample type validation | 1 day
  Establish if the hs-cTnI results obtained from finger prick capillary blood and fresh plasma are equivalent to results obtained for venous whole blood for the SpinChip hs-cTnI test when the analysis is performed by healthcare professionals. Equivalence between sample types will be evaluated using Bland Altman difference plots for evaluation of bias and regression analysis.

SECONDARY OUTCOMES:
Incidence of AEs, ADEs and DDs | 1 day
  Assess the safety of the SpinChip Platform, as measured by adverse events (AEs), adverse device effects (ADEs) and device deficiencies (DDs).

CONTACTS AND LOCATIONS:
Overall Officials: Helge Røsjø, MD/Professor, Principal Investigator — Akershus University Hospital, Akershus Clinical Research Center (ACR); Gro Leite Størvold, PhD, Study Director — SpinChip Diagnostics ASA
Locations (1):
- Akershus University hospital, Akershus Clinical Research Center (ACR), Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No